CLINICAL TRIAL: NCT03245684
Title: Assessment of the Inflammatory Response Associated With the Increase of Transpulmonary Pressure in Ipoxiemic Patients During Assisted Mechanical Ventilation
Brief Title: Assisted or Controlled Ventilation in Ards (Ascovent)
Acronym: ASCOVENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Alessandri, Dirigente medico I livello ( Medical Division of Anestesia andintensive care unit), University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCOVENT
Record Dates: First submitted 2017-08-04; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: ARDS; Ventilator-Induced Lung Injury; Mechanical Ventilation Complication; Inflammatory Response
Keywords: ARDS; Ventilator-induced Lung Injury; cytokines; mechanical ventilation
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure Support Ventilation (Experimental): after 48h of controlled ventilation the patient randomised in this arm will desedated and switched on Pressure Support Ventilation (PSV): patient's spontaneous activity will maintained and sedation will be maintained at a level of Richmond Assessment Sedation Scale (RASS) between -2 and -3. The level of pressure support (including PEEP) will be limited to ≤ 30 cmH2O; the pressure support level will ensure a tidal volume of 6 ml / Kg ideal body weight. PEEP, FiO2 and respiratory rate will be regulated according the ARDSnet protocol.
  assessment of inflammatory response during PSV
  Interventions: Diagnostic Test: assessment of inflammatory response during PSV
- Controlled Mechanical Ventilation (Active Comparator): patient's spontaneous activity will be shut done by sedation and/or respiratory muscles paralysis. Volume (during volume control) or pressure (during pressure control), PEEP, FiO2 and respiratory rate will be regulated according the ARDSnet protocol
  Interventions: Diagnostic Test: assessment of inflammatory response during PSV

INTERVENTIONS:
Diagnostic Test: assessment of inflammatory response during PSV — assessment cytokines level in BAL and plasma

SUMMARY:
The present pilot randomized controlled clinical trial will test the hypothesis that in patients with ARDS, fixing ventilator settings to the conventional protective ventilatory strategy (VT 6 ml/kg ideal body weight and Pplat ≤ 30 cmH2O, PEEP according the PEEP/FiO2 table), control modes of mechanical ventilation will be associated to a concentration of pulmonary and systemic inflammatory mediators lower than the concentration of inflammatory mediators observed during assisted modes of mechanical ventilation.

DETAILED DESCRIPTION:
All patients will be treated according to the sedation protocols and standards of care. Sedation will be guaranteed by continuous infusion of Propofol 2-4 ml / Kg / h, Remifentanil 0.05-0.1 mcg / Kg / min to obtain a RASS scale level of -5 of the RASS. Mio-resolution eventually obtained by a loading dose of 15 mg e.v. followed by a continuous infusion of 37.5 mg / h of besylated Cisatracury, will be reserved for patients with P/F <150.

During a 48 hrs pre-randomization period, control mechanical ventilation will be set with a Tidal Volume (VT) of 6 ml / kg (for ideal weight) and a Pplat limited to 30 cm H2O; inspiratory flow 50-70 l / min with end-of-breath pause of 0.2-0.5 sec, ratio I: E from 1: 1 to 1: 3, respiratory frequency of 20-35 steps to maintain 7.3 <pH <7.5. If the pH is <7.30 the respiratory frequency will increase up to 35 / min; If the pH is> 7.5, the respiratory rate will be progressively reduced to the target pH range. FiO2 and The PEEP will be set according to the ARDSnet table (33)

After 48 hours, the patient will be randomized through one of the following two groups:

Control Mechanical ventilation (CMV): patient's spontaneous activity will be shut done by sedation and/or respiratory muscles paralysis. Volume (during volume control) or pressure (during pressure control), PEEP, FiO2 and respiratory rate will be regulated according the ARDSnet protocol (33).

Pressure Support Ventilation (PSV): patient's spontaneous activity will maintained and sedation will be maintained at a level of Richmond Assessment Sedation Scale (RASS) between -2 and -3. The level of pressure support (including PEEP) will be limited to ≤ 30 cmH2O; the pressure support level will ensure a tidal volume of 6 ml / Kg ideal body weight. PEEP, FiO2 and respiratory rate will be regulated according the ARDSnet protocol (33)

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age who:

  1. Are intubated less than 24 hours since meeting the Berlin definition criteria for ARDS.
  2. Have a commitment to full support;
  3. Have no exclusion criteria

Exclusion Criteria:

1. Intubation and mechanical ventilation (any form) for > 24 hours;
2. Acute brain injury with Glasgow coma scale (GCS) <7;
3. Body mass index > 40;
4. Age < 18 years;
5. Neuromuscular disease that impairs ability to ventilate without assistance;
6. Severe chronic respiratory disease;
7. Burns > 40% total body surface area;
8. Malignancy or other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%;
9. Allogeneic bone marrow transplant within the last 5 years;
10. Chronic respiratory condition making patient respirator dependent;
11. Patient, surrogate, or physician not committed to full support;
12. Acute myocardial infarction or acute coronary syndrome within 30 days;
13. Moribund patient: not expected to survive 24 hours;
14. No consent/inability to obtain consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary concentration of inflammation mediators (broncho-alveolar lavage: BAL) | 96 hours
  Dosage of inflammatory mediators (tumor necrosis factor-α soluble receptors, interleukin-6, interleukin-8 and interleukin-1β and interleukin-1 receptor antagonist)

SECONDARY OUTCOMES:
Systemic concentration of inflammation mediators (plasma) | 96 hours
  The concentrations of the same mediators (tumor necrosis factor-α soluble receptors, interleukin-6, interleukin-8 and interleukin-1β and interleukin-1 receptor antagonist) in a sample of 10 ml of blood taken from a central venous line will be analyzed

OTHER OUTCOMES:
Number of ventilator-free days (VFDs) during the 28 days immediately after randomization | 28 days
Relationship between cytokine concentration and trans-pulmonary pressure | 96 hours
  End-expiratory and end-inspiratory occlusions will be performed. End-inspiratory Plateau Pressure. Pplat of the respiratory system (Pplatrs) will be the value of PAW after an end-inspiratory occlusion. End-inspiratory chest wall plateau pressure (PplatCW) will be measured as the variation in PES between end-expiratory and end-inspiratory occlusions; end-inspiratory plateau pressure of the lung (Pplatl) were estimated as Pplatrs - PplatCW

IPD SHARING:
Plan to Share IPD: Undecided